CLINICAL TRIAL: NCT03000049
Title: Bedside vs. Standard Microbiological Blood Culture Diagnostics - BEMIDIA Study
Acronym: BEMIDIA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Principal Investigator, Sven-Olaf Kuhn, Sven-Olaf Kuhn MD, University Medicine Greifswald
Other Study IDs: SD_BK_1_ANI
Record Dates: First submitted 2016-12-15; First posted 2016-12-21 (Estimated); Last update posted 2016-12-22 (Estimated); Status verified 2016-12

CONDITIONS: Sepsis Septic Shock
Keywords: sepsis; septic shock; blood cultures; anti-infective therapy
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: bedside blood culture

SUMMARY:
With a completely bedside blood culture diagnostics system (BACTEC blood culture system in combination with the Accelerate ID/AST System) it is possible to optimize the initial antimicrobial therapy in patients with sepsis and septic shock.

Prospective observational, open-label mono-center study to compare a completely bedside blood culture diagnostics system (BACTEC blood culture system in combination with the Accelerate ID/AST System and Curetis Univero System) with standard blood culture diagnostics in patients with sepsis or septic shock.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a new diagnosed sepsis or septic shock: emergency department, operating theatre, intensive care unit and planed blood culture diagnostics.
* informed written consent

Exclusion Criteria:

* Pediatric patients (< 18 Years)
* DNR-order

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with sepsis or septic shock with planned blood culture drawing
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-07 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Time to a significant change of antimicrobial therapy from the time of the diagnosis of sepsis or septic shock | Nov. 2016 - Nov. 2017

CONTACTS AND LOCATIONS:
Locations (1):
- Anesthesiology and Intensive Care Medicine Department, University of Greifswald, Germany, Greifswald, Germany

IPD SHARING:
Plan to Share IPD: No